CLINICAL TRIAL: NCT03025893
Title: A Phase II/III Study of High-dose, Intermittent Sunitinib in Patients With Recurrent Glioblastoma Multiforme: the STELLAR Study
Brief Title: A Phase II/III Study of High-dose, Intermittent Sunitinib in Patients With Recurrent Glioblastoma Multiforme
Acronym: STELLAR
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, M.E. van Linde, Medical Oncologist Department of Medical Oncology, Amsterdam UMC, location VUmc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016.221
Record Dates: First submitted 2017-01-09; First posted 2017-01-20 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Glioblastoma Multiforme; Glioblastoma, Adult; Glioblastoma; Recurrent Brain Tumor; GBM
Keywords: Sunitinib; Lomustine; High-dose; Intermittent
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Sunitinib; Lomustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sunitinib (Experimental): Patients in this experimental arm will receive sunitinib in a high-dose, intermittent schedule.
  Interventions: Drug: Sunitinib
- Lomustine (Active Comparator): Patients in this control arm will receive lomustine, currently used as second-line treatment in the case of recurrence.
  Interventions: Drug: Lomustine

INTERVENTIONS:
Drug: Sunitinib — Sunitinib, 300 mg administered orally in a weekly schedule.
  Other Names: Sutent
  Arms: Sunitinib
Drug: Lomustine — Lomustine 110 mg/m2, taken orally on day 1 every 6 weeks.
  Other Names: CCNU
  Arms: Lomustine

SUMMARY:
In this study the investigators will evaluate the effect of high-dose, intermittent sunitinib versus treatment with lomustine in patients with recurrent glioblastoma multiforme. The investigators hypothesize that sunitinib, when given in a high-dose, intermittent schedule, will achieve adequate concentration levels in the tumor and will, besides its anti-angiogenic properties, inhibit gliomagenesis by inhibition of multiple kinases.

DETAILED DESCRIPTION:
Study design: Multicenter, phase II/III, randomized clinical trial with high-dose sunitinib versus lomustine (CCNU) in patients with recurrent GBM.

Hypothesis: Sunitinib, when given in a high-dose, intermittent schedule, may exhibit improved efficacy in patients with recurrent GBM with an acceptable toxicity profile, compared to lomustine.

Study population: Adult patients with recurrent GBM.

Primary objective:

- To determine the effect of high-dose sunitinib versus lomustine on six-month progression-free survival (PFS6) in patients with recurrent GBM, using the RANO criteria.

Secondary objectives:

* To determine the effect of high-dose sunitinib on overall survival (OS 9, OS 12) in patients with recurrent GBM.
* To assess the objective radiological response rate, using the RANO criteria.
* To assess toxicity, using the Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0.
* To assess patient-oriented criteria: steroid use and health-related quality of life (reported by patients and caregivers/relatives).
* To explore the potential value of blood markers for molecular diagnostics, disease and response monitoring.
* To explore if MGMT promoter methylation status modulates the response to sunitinib.

Treatment: After randomization, 100 patients will be divided equally over two treatment groups and will receive:

* Group 1 (experimental arm): Sunitinib, 700 mg administered orally every 2 weeks.
* Group 2 (control arm): Lomustine 110 mg/m2, taken orally on day 1 every 6 weeks.

Disease will be assessed by MRI according to an uniform neuro-oncology protocol every 6 weeks for the first 6 months and every 12 weeks until documented progression. Safety profile of both treatment strategies will be assessed separately for each cycle of therapy and every 12 weeks after the end of treatment if adverse effects have not resolved or are newly emerging. Furthermore, quality of life assessment takes place every 6 weeks using questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Signed (by the patient or legally acceptable representative) and dated Informed Consent Form
2. Histologically confirmed de novo or secondary glioblastoma with unequivocal first progression, at least 3 months off radiotherapy.
3. No more than one line of chemotherapy (concurrent and adjuvant temozolomide based chemotherapy including in combination with another investigational agent is considered one line of chemotherapy). Chemotherapy must have been completed at least 4 weeks prior to randomization.
4. Patients may have undergone surgery for recurrence. If operated, residual and measurable disease after surgery is not required but surgery must have confirmed the recurrence.
5. No radiotherapy, stereotactic radiosurgery or brachytherapy as treatment for recurrence.
6. Patients must have a Karnofsky Performance Score ≥ 70%
7. Patients need to have adequate hematological, renal and hepatic function as assessed by the following laboratory requirements to be conducted within seven days prior to start study treatment:

   1. Hemoglobin ≥ 7.0 mmol/L
   2. Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   3. Platelet count ≥ 100 x 109/L
   4. ALAT and ASAT ≤ 2.5 x ULN
   5. Serum creatinine eGFR ≥ 50 ml/min
   6. Albumin ≥ 25 g/L
8. Age ≥ 18 years

Exclusion Criteria:

1. Evidence of a significant uncontrolled concomitant disease, such as cardiovascular disease (including stroke, New York Heart Association Class III or IV cardiac disease or myocardial infarction within 6 months prior to screening, unstable arrhythmia, clinically significant valvular heart disease and unstable angina); nervous system, pulmonary (including obstructive pulmonary disease and history of symptomatic bronchospasm), renal, hepatic, endocrine, or gastrointestinal disorders; or a serious non-healing wound or fracture.
2. Patients with a prior (< 5 years) or concomitant second malignancy.
3. Prior radiotherapy in the abdomen or in the lungs or in more than 3 vertebrae in the spine (Less than 3 vertebrae are considered a small radiation field and eligibility will be decided on an individual basis from the PI).
4. Poorly controlled hypertension despite adequate blood pressure medication. Blood pressure must be ≤ 160/95 mmHg at the time of screening on a stable antihypertensive regimen. Blood pressure must be stable on at least 2 separate measurements.
5. Known active bacterial, viral, fungal, mycobacterial, or other infection (including HIV and atypical mycobacterial disease, but excluding fungal infection of the nail beds.)
6. Initial MR-scan of the brain showing intratumoral hemorrhage, except for stable post-operative grade 1 hemorrhage.
7. Known hypersensitivity to sunitinib or to its excipients.
8. Presence of any significant central nervous system or psychiatric disorder(s) that would interfere with the patient's compliance.
9. Use of full-dose oral or parenteral anticoagulants or thrombolytic agent for therapeutic (as opposed to prophylactic) purposes.
10. Use of strong hepatic enzyme-inducing antiepileptic drugs, such as carbamazepine, phenobarbital and phenytoin. If a patient uses one or more of these specific antiepileptic drugs, they must switch to an antiepileptic drug that does not interact with cytochrome P450 (CYP450) liver enzymes, such as levetiracetam, prior to the start of study treatment.
11. Drug or alcohol abuse.
12. Females who are pregnant or breast-feeding.
13. Any evidence of a disease or condition that might affect compliance with the protocol or interpretation of the study results or render the patient at high risk from treatment complications.
14. Unwillingness or inability to comply with study and follow-up procedures.
15. Clinically significant history of liver disease, including viral or other hepatitis, current alcohol abuse, or cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-31 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Six-month progression-free survival (PFS-6) | From the date of randomization up to the date of first progression or death (any cause) whichever comes first, assessed up to 36 months (End of Study).

SECONDARY OUTCOMES:
Overall survival (OS) | From the date of randomization up to the date of death, assessed up to 36 months. If study medication is discontinued for any reason, survival follow-up takes place every 12 weeks, also assessed up to 36 months (End of Study).
Objective radiological response rate | Disease will be assessed by MRI every 6 weeks for the first 6 months and every 12 weeks until documented progression, assessed up to 36 months (End of Study).
  Response will be assessed according to the RANO criteria.
Adverse events (AEs) | AEs will be monitored at every visit during study treatment or after discontinuation of study treatment in the case adverse events have not subsided, assessed up to 36 months (End of Study).
  At the end of the study, after 36 months, the number of participants with adverse events that are related to both treatments will be assessed and compared.
Health-related quality of life (HRQoL) | HRQoL assessments will be performed at baseline and every 6 weeks until documented progression, assessed up to 36 months (End of Study).
  Steroid use will be documented at every treatment cycle as an objective parameter for HRQoL. Furthermore, HRQoL will also be measured via EORTC questionnaires, which will be filled in by the participants every 6 weeks BEFORE their MRI.
Blood markers (TEP: tumor educated platelets, and miRNA) | Blood samples for RNA profiling will be drawn simultaneously with regular blood samples on five specific time points during study treatment and will be assessed after 36 months (End of Study).
  The five specific time points during study treatment are: (1) at baseline; (2) at the first outpatient visit; (3) after two weeks of treatment; (4) at the first response evaluation (first MRI); and (5) at the time of progression.
MGMT promoter methylation status | At the end of the study (after 36 months), the treatment outcomes of all patients will be correlated with the MGMT promoter methylation status.
  Previously obtained resection or biopsy material from the first-line treatment of these participants will be requested at the time of inclusion and used to determine the MGMT methylation status. After the End of Study (after 36 months) the MGMT promoter methylation status will be correlated with the response to treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Myra E Van Linde, MD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (3):
- Netherlands (3):
  - VU University Medical Center, Amsterdam
  - University Medical Center Groningen, Groningen
  - Radboud UMC, Nijmegen